CLINICAL TRIAL: NCT00002716
Title: PHASE III STUDY OF HEPATIC ARTERY FLOXURIDINE (FUDR), LEUCOVORIN (LV), AND DEXAMETHASONE (DEX) VERSUS SYSTEMIC 5-FLUOROURACIL (5-FU) AND LEUCOVORIN (LV) AS TREATMENT FOR HEPATIC METASTASES FROM COLORECTAL CANCER
Brief Title: Combination Chemotherapy in Treating Patients With Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9481; U10CA031946 (NIH); CDR0000064553 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Dexamethasone; Floxuridine; Fluorouracil; Leucovorin; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I - laparotomy + conventional surgery + chemotherapy (Experimental): Patients undergo laparotomy for placement of a hepatic artery catheter and then subcutaneous placement of a hepatic artery infusion pump. Patients with unresected primary disease also undergo resection at the time of catheter and pump placement. Beginning within 1-2 weeks after surgery, patients receive floxuridine, dexamethasone, and leucovorin calcium (CF) via continuous hepatic artery infusion on days 1-14. Treatment for patients continues every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Quality of life and medical resource utilization are assessed at baseline, every 3 months for 1 year, and then at 18 months.
  Patients are followed every 3 months.
  Interventions: Drug: dexamethasone; Drug: floxuridine; Drug: leucovorin calcium; Procedure: laparotomy; Procedure: conventional surgery
- Arm II - conventional surgery + chemotherapy (Experimental): Patients receive CF IV and fluorouracil IV on days 1-5. Patients with unresected primary disease undergo resection within 3-4 weeks before initiation of chemotherapy.
  Treatment for patients continues every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Quality of life and medical resource utilization are assessed at baseline, every 3 months for 1 year, and then at 18 months.
  Patients are followed every 3 months.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Procedure: conventional surgery

INTERVENTIONS:
Drug: dexamethasone
  Arms: Arm I - laparotomy + conventional surgery + chemotherapy
Drug: floxuridine
  Arms: Arm I - laparotomy + conventional surgery + chemotherapy
Drug: fluorouracil
  Arms: Arm II - conventional surgery + chemotherapy
Drug: leucovorin calcium
Procedure: laparotomy
  Arms: Arm I - laparotomy + conventional surgery + chemotherapy
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which chemotherapy regimen is more effective for metastatic colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of intrahepatic floxuridine, leucovorin, and dexamethasone with that of systemic fluorouracil and leucovorin in treating patients who have unresectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy, toxicity, and cost of hepatic artery infusion of floxuridine, leucovorin calcium (CF), and dexamethasone vs IV fluorouracil and IV CF after resection of primary disease in patients with hepatic metastases secondary to colorectal cancer.
* Compare the quality of life of patients treated with these regimens.
* Measure the level of thymidylate synthase present in liver metastases, and correlate these levels with objective response and survival in patients treated with these regimens.
* Assess the p53 mutations, and correlate findings with objective response and survival in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, percentage of liver involvement on CT scan or MRI (less than 30% vs 30% to under 70%), prior chemotherapy (none vs adjuvant chemotherapy comprising fluorouracil (5-FU) and leucovorin calcium (CF) or 5-FU, CF, and levamisole (LEV) completed at least 1 year before study vs adjuvant chemotherapy comprising 5-FU with or without LEV completed at least 6 months before study), and synchronous disease (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Unresectable liver metastases secondary to colorectal cancer

  * Less than 70% liver involvement on CT scan or MRI
  * Liver biopsy required before study unless 1 of the following conditions are met:

    * Carcinoembryonic antigen greater than 30
    * 5 or more liver metastases visible on CT scan or MRI
    * Greater than 50% to under 70% liver involvement on CT scan or MRI
* Histologically proven primary colorectal cancer that is resected or appears resectable on CT scan and physical exam

  * Documentation of previously resected primaries must be based on pathologic results of the resected tumor
  * Histological documentation of synchronous disease must be based on 1 of the following:

    * Biopsy of primary colorectal tumor before study
    * Suspicious lesion on barium enema, colonoscopy, or sigmoidoscopy, and a liver biopsy positive for adenocarcinoma consistent with the primary colorectal tumor
* Measurable disease

  * Clearly defined liver mass measuring at least 2 cm or at least 3 liver masses on CT scan or MRI
* No evidence of extrahepatic disease on CT scan and physical exam
* No portal vein occlusion or ascites

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Hepatic:

* Bilirubin no greater than 2 times normal

Other:

* No other malignancy within the past 5 years except inactive nonmelanomatous skin cancer, carcinoma in situ of the cervix, or grade 1 bladder cancer
* Not pregnant or nursing
* Fertile patients must use effective contraception

Chemotherapy:

* At least 1 year since prior adjuvant chemotherapy comprising fluorouracil (5-FU) and leucovorin calcium (CF) or 5-FU, CF, and levamisole (LEV)
* At least 6 months since prior adjuvant chemotherapy comprising 5-FU with or without LEV
* No other prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except for nondisease-related conditions, e.g.:

  * Steroids for adrenal failure
  * Insulin for diabetes
  * Intermittent dexamethasone as an antiemetic

Radiotherapy:

* No prior radiotherapy to the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 1996-01; Primary Completion 2006-03 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
Time to progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Kemeny, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (14):
- United States (11):
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - MetroHealth Medical Center, Cleveland, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Kemeny NE, Niedzwiecki D, Hollis DR, Lenz HJ, Warren RS, Naughton MJ, Weeks JC, Sigurdson ER, Herndon JE 2nd, Zhang C, Mayer RJ. Hepatic arterial infusion versus systemic therapy for hepatic metastases from colorectal cancer: a randomized trial of efficacy, quality of life, and molecular markers (CALGB 9481). J Clin Oncol. 2006 Mar 20;24(9):1395-403. doi: 10.1200/JCO.2005.03.8166. Epub 2006 Feb 27. PMID 16505413
- [Result] Kemeny NE, Niedzwiecki D, Hollis DR, et al.: Final analysis of hepatic arterial infusion (HAI) versus systemic therapy for hepatic metastases from colorectal cancer: a CALGB randomized trial of efficacy, quality of life (QOL), cost effectiveness, and molecular markers. [Abstract] American Society of Clinical Oncology 2005 Gastrointestinal Cancers Symposium, 27-29 January 2005, Miami, Florida. A-183, 2005.
- [Result] Mandola MV, Stoehlmacher J, Muller-Weeks S, Cesarone G, Yu MC, Lenz HJ, Ladner RD. A novel single nucleotide polymorphism within the 5' tandem repeat polymorphism of the thymidylate synthase gene abolishes USF-1 binding and alters transcriptional activity. Cancer Res. 2003 Jun 1;63(11):2898-904. PMID 12782596
- [Result] Pullarkat ST, Stoehlmacher J, Ghaderi V, Xiong YP, Ingles SA, Sherrod A, Warren R, Tsao-Wei D, Groshen S, Lenz HJ. Thymidylate synthase gene polymorphism determines response and toxicity of 5-FU chemotherapy. Pharmacogenomics J. 2001;1(1):65-70. doi: 10.1038/sj.tpj.6500012. PMID 11913730